CLINICAL TRIAL: NCT00751530
Title: Outcomes of Early Raltegravir Experience: Comparison of Virologic Response in Regimens Not Containing a Protease Inhibitor in the Antiretroviral Background Regimen Versus a Protease Inhibitor in the Background Regimen
Brief Title: BRAVO: Background Regimen of Raltegravir on Virologic Outcome
Acronym: BRAVO
Status: Completed | Type: Observational
Sponsor: Community Research Initiative of New England (Other)
Responsible Party: Sponsor
Other Study IDs: 07-11
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Results first posted 2011-06-17 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-07

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; raltegravir; BRAVO; protease inhibitor; treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Protease Inhibitor Group: Subjects who required a protease inhibitor in their new ART regimen
  Interventions: Drug: raltegravir
- Non-protease Inhibitor: Subjects who did not take a protease inhibitor in their regimen
  Interventions: Drug: raltegravir

INTERVENTIONS:
Drug: raltegravir — New combination ART incorporating raltegravir with other ARVs.

SUMMARY:
This is a retrospective chart review of participants in raltegravir expanded access program and will compare virologic response in regimens not containing a protease inhibitor in the antiretroviral background regimen to regimens containing a protease inhibitor in the background regimen.

DETAILED DESCRIPTION:
EAP charts from patients at the study sites who meet the inclusion criteria will be reviewed and data abstracted. A comparison of the response to treatment by viral load measurement with raltegravir will be compared in patients whose regimens contained a protease inhibitor (PI) with those that did not contain a PI. Other endpoints will also be assessed including percent of patients with viral loads less than 400 copies/ml, less than 50 copies/ ml, CD4 cell changes, consequences of failure of raltegravir and use of predictive parameters such as GSS and PSS.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously enrolled in the MK 0518 EAP are eligible
* Patients not enrolled in the MK 0518 EAP (or other Raltegravir protocols) but who meet the specific EAP protocol entry criteria are eligible:

  * Age >= 16 years
  * Limited or no treatment options due to resistance or intolerance to multiple antiretroviral regimens, documented resistance to at least one drug in each of the 3 classes of oral ARTs (NRTI, NNRTI, PI) by genotype or phenotype testing, intolerance defined as having had a clinically significant adverse event which in the opinion of the clinician provides a contraindication to the use of any drug in that class iii. Patient did not achieve virologic suppression on ART regimen prior to receipt of raltegravir iv. Patient was clinically stable at time of initiation of raltegravir, eg. clinical status and all chronic medications (except ARTs) unchanged for >= 2 weeks prior to raltegravir receipt.
* Patient received raltegravir for at least 8 weeks
* Baseline and week 8 or later HIV viral load done and available for review
* Resistance test (either genotypic or phenotypic test) available prior to receipt of raltegravir

Exclusion Criteria:

* Patient did not receive approved raltegravir dose of 400 mg BID for at least 8 weeks.
* Patient chart not available for review.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of individuals who were previously enrolled in raltegravir expanded access program(EAP) and completed at least 8 weeks of treatment with raltegravir, whose chart from EAP program is available for review, and whose resistance testing prior to initiation of raltegravir is available.
Sampling Method: Non-Probability Sample
Enrollment: 442 (Actual)
Dates: Start 2008-03-01 (Actual); Primary Completion 2009-06-15 (Actual); Study Completion 2009-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Skiest, MD, Principal Investigator — Community Research Initiative
Locations (15):
- United States (15):
  - Light Source Medical, Los Angeles, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - Synergy Hematology and Oncology, Los Angeles, California
  - Quest Clinical Research, San Francisco, California
  - Connecticut Health Care Group, Glastonbury, Connecticut
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Capital Medical Associates PC, Washington D.C., District of Columbia
  - Orlando Immunology Center, Orlando, Florida
  - Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Community Research Initiative, Boston, Massachusetts
  - Community Research Initiative - West, Springfield, Massachusetts
  - Infectious Diseases and HIV Medicine Immunodeficiency Clinic, Buffalo, New York
  - Bellman, MD, New York, New York
  - Mounzer, MD, Philadelphia, Pennsylvania
  - Dr. Nicholaos C. Bellos & Associates, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Protease Inhibitor Group | Non-protease Inhibitor
Started | 332 | 110
Completed | 332 | 110
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Protease Inhibitor Group | Non-protease Inhibitor | Total
Number analyzed (Participants) | 254 | 86 | 340
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 247 | 82 | 329
  >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 13 | 38
  Male | 229 | 73 | 302
Region of Enrollment [Number; unit: participants]
  United States | 254 | 86 | 340

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With Viral Load < 75 Copies/ mL at Week 12
Description: The HIV RNA (viral load) was measured using standard of care testing via local laboratories.
Time Frame: 12 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | Protease Inhibitor Group | Non-protease Inhibitor
Number analyzed (Participants) | 254 | 86
Percentage of participants | 84 | 86

2. Secondary Outcome: CD4 Cell Changes Among Participants in PI vs Non-PI Group
Description: CD4 cell counts were measured using standard of care testing via local laboratories.
Time Frame: baseline to 24 Weeks
Measure: Mean (Full Range); unit: cells/mm3
Arm/Group | Protease Inhibitor Group | Non-protease Inhibitor
Number analyzed (Participants) | 129 | 44
cells/mm3 | -96.6 (NA) [-310 to 768] | -134.8 (NA) [-385 to 42]

3. Secondary Outcome: Baseline Genotypic Sensitivity Score (GSS). The Minimal Value Was 0 and the Maximum Values Was 5.4. (0 = Minimal to no Activity in Regimen and 5.4 = High to Maximal Activity in Regimen)
Description: The baseline GSS is calculated by the sum of resistance scores for each drug in the regimen. For each drug in the regimen a resistance score of 0, 0.5 or 1 was assigned for high, low or no levels of resistance, respectfully. The resistance assignment was based on either the Stanford database interpretation or presence of primary IAS mutation levels of resistance. Inclusion of maraviroc or new use of enfuvirtide in the regimen was scored a 1.0. The sum of the scores of the active drugs, not including raltegravir, constituted the baseline GSS.
Time Frame: Baseline
Measure: Mean (Full Range); unit: score
Arm/Group | Protease Inhibitor Group | Non-protease Inhibitor
Number analyzed (Participants) | 254 | 86
score | 1.8 [0 to 5.4] | 1.7 [0 to 3.5]

4. Primary Outcome: Percentage of Participants With Viral Load < 400 Copies /mL at Week 12.
Description: The HIV RNA (viral load) was measured using standard of care testing via local laboratories.
Time Frame: 12 Weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | Protease Inhibitor Group | Non-protease Inhibitor
Number analyzed (Participants) | 254 | 86
Percentage of Participants | 84 | 86

5. Secondary Outcome: Percentage of Participants Using Etravirine in Background Regimen
Description: These results report the percent of participants using Etravirine in the background regimen.
Time Frame: Background regimen (no specific time frame)
Measure: Number; unit: Percentage of Participants
Arm/Group | Protease Inhibitor Group | Non-protease Inhibitor
Number analyzed (Participants) | 100 | 58
Percentage of Participants | 33 | 58

ADVERSE EVENTS:
Arm/Group | Protease Inhibitor Group | Non-protease Inhibitor
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site Investigators (PIs) agree not to individually publish the results of the study. They may participate in a joint publication of the study results with the sponsor.